CLINICAL TRIAL: NCT05862961
Title: Towards a Better Classification of Respiratory Amyloidosis. Contribution of Proteomic Analysis Based on Tandem Mass Spectrometry
Brief Title: Better Classification of Respiratory Amyloidosis
Acronym: B-AR
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220270
Record Dates: First submitted 2023-03-27; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-03

CONDITIONS: Amyloidosis
Keywords: respiratory amyloidosis; proteomic analysis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — fixed tissue (Lung biopsy, Bronchial biopsy; trans-thoracic lung biopsy, trans-bronchial lung biopsy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The B-AR project is based on a retrospective analysis of amyloidosis typing and the identification of their amylogenic protein.This work should be able to unite many clinicians, including pulmonologists and pathologists around a rare disease that still suffers from insufficient data.

DETAILED DESCRIPTION:
The B-AR study will highlight the interest of proteomic analysis of amyloidosis compared to their identification by immunostaining. The objective is to reduce diagnostic wandering and to improve patient management. The typing of respiratory amyloidosis will allow a better characterization of the disease and thus, to propose a dedicated therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > to 18 years with amyloidosis on a histological sample of the tracheobronchial or pulmonary tree.

Exclusion Criteria:

* Subject receiving state medical aid
* Subject deprived of freedom, or under a legal protective measure (example: patients under guardianship or curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with respiratory amyloidosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Number of cases with identification of the amylogenic protein in respiratory amyloidosis. | 1 day (at inclusion)
  Identification of amylogenic protein by Proteomic Analysis Based on Tandem Mass Spectrometry on histological sample of the tracheobronchial or pulmonary tree.

SECONDARY OUTCOMES:
Distribution and severity of amyloidosis | 1 day (at inclusion)
  association between typing and respiratory involvement

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagül UZUNHAN, Pr,MD, PhD, Study Director — APHP Hôpital Avicenne